CLINICAL TRIAL: NCT04516538
Title: Effects of Mode of Contraction on Neuromuscular Fatigue in Young People Aged 18 to 35, Aged 60 to 80 and Very Old People Aged Over 80
Brief Title: Effects of Mode of Contraction on Neuromuscular Fatigue
Acronym: DYN-AGING
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19CH178; 2020-A00016-33 (Other: ANSM)
Record Dates: First submitted 2020-07-29; First posted 2020-08-18 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Volunteers
Keywords: Aging; neuromuscular performance; central fatigue; peripheral fatigue; dynamic
MeSH Terms: interventions — Mental Status and Dementia Tests; Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Young people (Experimental): Men or Women under 35 years old
  Interventions: Diagnostic Test: 6 Minutes Walk Test; Diagnostic Test: Timed up and go; Diagnostic Test: Isokinetic Body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Cycloergometer body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Isometric BW-QIF Test (Body weight-based quadriceps intermittent fatigue test)
- Old people (Experimental): Men or Women between 60 and 80 years old
  Interventions: Diagnostic Test: 6 Minutes Walk Test; Diagnostic Test: Timed up and go; Diagnostic Test: Isokinetic Body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Cycloergometer body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Isometric BW-QIF Test (Body weight-based quadriceps intermittent fatigue test)
- Very old people (Experimental): Men or Women over 80 years old
  Interventions: Behavioral: Mini Mental State Examination; Diagnostic Test: 6 Minutes Walk Test; Diagnostic Test: Timed up and go; Diagnostic Test: Isokinetic Body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Cycloergometer body weight-based quadriceps intermittent fatigue test (BW-QIF Test); Diagnostic Test: Isometric BW-QIF Test (Body weight-based quadriceps intermittent fatigue test)

INTERVENTIONS:
Behavioral: Mini Mental State Examination — test for evaluating a person's cognitive functions and memory capacity
  Arms: Very old people
Diagnostic Test: 6 Minutes Walk Test — a standardized test of an individual's functional ability that involves walking the greatest distance a person can walk in six minutes. This walking may be limited by shortness of breath or fatigability.
Diagnostic Test: Timed up and go — A simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time it takes for a person to get up from a chair, walk three metres, turn around, walk to the chair and sit down.
Diagnostic Test: Isokinetic Body weight-based quadriceps intermittent fatigue test (BW-QIF Test) — The BW-QIF test is an interval incremental contraction test including blocks of discontinuous 100-s effort. Neuromuscular evaluation of the knee extensors between blocks (duration 25 s) includes one maximal voluntary contraction, one contraction at the 60% of the actual maximal force and at the 80% of the actual maximal force. During each contraction, transcranial magnetic stimulation over the motor cortex will be delivered to assess corticospinal voluntary activation (central fatigue). Single-twitch electrical stimulations will be delivered on the femoral nerve during the maximal voluntary contraction and at rest to evaluate peripheral fatigue.
  The isokinetic BW-QIF test blocks consist in 100 contractions at 120° deg.s-1 and 60° of range of motion (0.5-s contraction /0.5-s rest).
Diagnostic Test: Cycloergometer body weight-based quadriceps intermittent fatigue test (BW-QIF Test) — The BW-QIF test is an interval incremental contraction test including blocks of discontinuous 100-s effort. Neuromuscular evaluation of the knee extensors between blocks (duration 25 s) includes one maximal voluntary contraction, one contraction at the 60% of the actual maximal force and at the 80% of the actual maximal force. During each contraction, transcranial magnetic stimulation over the motor cortex will be delivered to assess corticospinal voluntary activation (central fatigue). Single-twitch electrical stimulations will be delivered on the femoral nerve during the maximal voluntary contraction and at rest to evaluate peripheral fatigue.
  The BW-QIF test blocks on the cycloergometer consist in 100 s of cycling at 60 Revolution Per Minute (RPM).
Diagnostic Test: Isometric BW-QIF Test (Body weight-based quadriceps intermittent fatigue test) — The BW-QIF test is an interval incremental contraction test including blocks of discontinuous 100-s effort. Neuromuscular evaluation of the knee extensors between blocks (duration 25 s) includes one maximal voluntary contraction, one contraction at the 60% of the actual maximal force and at the 80% of the actual maximal force. During each contraction, transcranial magnetic stimulation over the motor cortex will be delivered to assess corticospinal voluntary activation (central fatigue). Single-twitch electrical stimulations will be delivered on the femoral nerve during the maximal voluntary contraction and at rest to evaluate peripheral fatigue.
  The isometric BW-QIF test blocks consist in 10 contractions (5-s contraction / 5-s rest).

SUMMARY:
Aging is associated with multiple deteriorations of the neuromuscular system. Given the increase in life expectancy, the investigators can now distinguish old adults (>60 years old) who conserve their neuromuscular capacities with regular physical activity and very old adults (>80 years old) who suffer from an inexorable decline, even if the number of octogenarians and their quality of life are progressively increasing. However, the most part of the literature on fatigue and neuromuscular capacity with aging focused on isometric tasks. The results showed a significant decrease in maximal force production capacity and a greater resistance to fatigue for old people compared to the young population. When fatigue is induced trough dynamic contractions, greater fatigability was observed in old adults compared to young adults. Investigations performed on the population aged over 80 years old are rare, showing greater fatigability in octogenarians than old men (aged 60-80 years old) during isometric tasks. The knowledge about the effects of dynamic contractions in this population are limited, and performed uniquely in single leg isokinetic mode. Evaluations that require the use of both legs and higher muscle mass involved in the task (cycloergometer) are needed. Understanding neuromuscular fatigue and fatigability across different exercise modalities is necessary to set adapted physical activity programs aimed to maintain autonomy in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Belong to a defined age group: young (18 to 35 years old inclusive), old (60 to 80 years old inclusive) and very old (81 to 95 years old inclusive),
* Signed written consent form
* Being affiliated to social security

Exclusion Criteria:

* Pathology or surgery resulting in a locomotor disorder, within 6 months prior to the study,
* Chronic neurological, motor or psychological pathologies
* Use of neuro-active substances likely to alter cortico-spinal excitability (hypnotics, antiepileptics, psychotropic drugs, muscle relaxants) for the duration of the study.
* Contraindication to magnetic stimulation:
* Cardiac or respiratory insufficiency.
* Cardiac pacemaker.
* Cardiac valve wear and serious cardiovascular diseases.
* Presence of prosthetic material or ferromagnetic foreign bodies in the head.
* Presence of cochlear implants or ocular prosthetic material.
* History of neurosurgical interventions.
* Neurological diseases that may affect brain structures and cognitive abilities (e.g., intracranial tumour, multiple sclerosis, history of stroke or traumatic brain injury).
* History of comitiality, contralateral knee pathology or pathology of the musculoskeletal system.
* Mini Mental State Examination < 20

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Maximum Voluntary Contraction (%) - all participants | Immediately after pedalling on an ergocycle
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.

SECONDARY OUTCOMES:
Percentage of Maximum Voluntary Contraction (%) - 18-35 years old participants | Before and immediately after pedalling on an ergocycle
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - 60-80 years old participants | Before and immediately after pedalling on an ergocycle
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - more than 80 years old participants | Before and immediately after pedalling on an ergocycle
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - more than 80 years old participants | Before and immediately after isometric contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - 60-80 years old participants | Before and immediately after isometric contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - 18-35 years old participants | Before and immediately after isometric contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - 18-35 years old participants | Before and immediately after concentric isokinetic contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - 60-80 years old participants | Before and immediately after concentric isokinetic contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.
Percentage of Maximum Voluntary Contraction (%) - more than 80 years old participants | Before and immediately after concentric isokinetic contractions
  The measurement of the maximum voluntary contraction is carried out at rest with the instruction to contract the extensor muscles of the knee as hard as possible by pushing against a fixed pedal. This force is measured by an isokinetic ergometer.

OTHER OUTCOMES:
Percentage of voluntary activation (%) | Before and immediately after concentric isokinetic contractions
  To compare voluntary Activation of the extensor muscles of the knee by peripheral nerve stimulation between 18-35 years old, 60-80 years old and more than 80 years old participants.
Percentage of voluntary activation (%) | Before and immediately after isometric contractions
  To compare voluntary Activation of the extensor muscles of the knee by peripheral nerve stimulation between 18-35 years old, 60-80 years old and more than 80 years old participants.
Percentage of voluntary activation (%) | Before and immediately after pedalling on an ergocycle
  To compare voluntary Activation of the extensor muscles of the knee by peripheral nerve stimulation between 18-35 years old, 60-80 years old and more than 80 years old participants.
Difference in amplitude of electric shock at rest (% of shock) | Before and immediately after pedalling on an ergocycle
  To compare the amplitude of the electric shock at rest of the extensor muscles of the knee between 18-35 years old, 60-80 years old and more than 80 years old participants.
Difference in amplitude of electric shock at rest (% of shock) | Before and immediately after isometric contractions
  To compare the amplitude of the electric shock at rest of the extensor muscles of the knee between 18-35 years old, 60-80 years old and more than 80 years old participants.
Difference in amplitude of electric shock at rest (% of shock) | Before and immediately after concentric isokinetic contractions
  To compare the amplitude of the electric shock at rest of the extensor muscles of the knee between 18-35 years old, 60-80 years old and more than 80 years old participants.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luneau E, Rozand V, Rimaud D, Foschia C, Millet GY. Walking Economy and Preferred Speed in Old and Very Old Men. Med Sci Sports Exerc. 2025 Feb 1;57(2):400-412. doi: 10.1249/MSS.0000000000003565. Epub 2024 Sep 17. PMID 39285590
- [Derived] Varesco G, Luneau E, Millet GY, Feasson L, Lapole T, Rozand V. Age-Related Differences between Old and Very Old Men in Performance and Fatigability Are Evident after Cycling but Not Isometric or Concentric Single-Limb Tasks. Med Sci Sports Exerc. 2023 Sep 1;55(9):1641-1650. doi: 10.1249/MSS.0000000000003181. Epub 2023 Apr 4. PMID 37580874